CLINICAL TRIAL: NCT00588185
Title: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone Pet Imaging in Patients With Progressive Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00-095
Record Dates: First submitted 2007-12-26; First posted 2008-01-08 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
Keywords: Progressive Prostate Cancer; [18F]-Fluoro-2-Deoxy-D-Glucose; [18F] Dihydro-Testosterone; Pet Imaging; Pet scan; 00-095
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone
  Interventions: Drug: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone

INTERVENTIONS:
Drug: [18F]-Fluoro-2-Deoxy-D-Glucose and -[18F] Dihydro-Testosterone — Registered patients will undergo PET scanning using either FDHT alone or FDG and FDHT depending on the clinical question being asked. Scans will be performed serially at baseline, week 4, week 12, and every 12 weeks of treatment up to a maximum of 8 FDHT/FDG scan set in a 12 month period (maximum 40 scan sets per lifetime) unless the therapeutic protocol or scientific rationale of the therapeutic drug being applied specifically dictates an alternative schedule. Patients may have blood drawn for the purposes of establishing the pharmacokinetics of FDHT and may also undergo an initial dynamic scan if further pharmacokinetic information is warranted, followed by a standard whole body image. If no further pharmacokinetic information is warranted, then patients will only undergo a standard whole body image.

SUMMARY:
This study will use PET scans, which is a type of x-ray test that uses a radiotracer, to see whether these scans may be better able to find places in the body where your prostate cancer may have spread.

DETAILED DESCRIPTION:
Our preliminary studies have shown that whole body FDG-PET imaging identifies areas of abnormal metabolism in a majority of tumor sites in patients with progressive disease and that changes in FDG accumulation parallel changes in PSA after treatment. This suggests that changes in FDG metabolism may provide an early assessment of treatment outcomes. In previous work we established a methodology to examine a radiotracer in patients with progressive disease and abnormal imaging studies, which we have applied to the clinical states of non-castrate and castrate metastatic disease. This design is characterized by:

1) Evaluation of uptake on a site-by-site basis in relation to conventional studies 2) Standardization of uptake values in tumor relative to a normal organ 3) Controlling for progression using standard measures of progression including a rising PSA, new or enlarging lesions on bone or transaxial imaging, and new symptoms of disease. In the present study we are evaluating fluorinated dihydrotestosterone (FDHT) in addition to FDG. FDHT is targeted to the AR and has been shown in preliminary studies to visualize prostate cancers in man. This study will apply our established methods to investigate FDHT imaging in patients with progressive prostate cancer. In the selected cases where tumor is available, we will study associations between FDHT accumulation and AR expression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed prostate cancer.
* Progressive disease manifest by either:
* Imaging modalities:
* Bone Imaging: New osseous lesions on bone imaging (bone scintigraphy or NaF PET scan) and/or MRI or CT: An increase in measurable soft tissue disease, or the appearance of new sites of disease. Or
* Biochemical progression: A minimum of three rising PSA values from a baseline that are obtained 1 week or more apart, or 2 measurements 2 or more weeks apart.
* Visible lesions by either CT, bone imaging, or MRI consistent with disease.
* Informed consent.

Exclusion Criteria:

* Previous anaphylactic reaction to either FDHT or FDG
* Hepatic: Bilirubin > 1.5 x upper limit of normal (ULN), AST/ALT >2.5 x ULN, albumin < 2 g/dl, and GGT > 2.5 x ULN IF Alkaline phosphatase > 2.5 x ULN
* Renal: Creatinine >1.5 x ULN or creatinine clearance < 60 mL/min

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To study the accumulation and biodistribution of FDHT in patients with progressive prostate cancer. The accumulation and location of FDHT activity will be assessed on a site by site basis and correlated with radionuclide bone scan, CT and MRI. | Baseline, 4 weeks and 12 weeks

SECONDARY OUTCOMES:
The kinetics, metabolism, and biodistribution will be assessed. | Baseline. 4 weeks and 12 weeks
To correlate the accumulation of 18FDHT to 18FDG. | 2 years
To study changes in 18FDHT accumulation over time in patients treated with: Castration and other hormones, Chemotherapy, Agents directed toward the androgen receptor | 2 years
relationship between FDHT uptake and tumor diffusivity | 2 years
  assessed by MRI.
relationship between FDHT uptake and tissue analyses | 2 years
  of AR expression

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, M.D., Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org